CLINICAL TRIAL: NCT05554523
Title: How Does Skin Tone Affect Quantitative Photoacoustic Imaging
Acronym: PAISKINTONE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cambridge (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Principal Investigator, Sarah Bohndiek, Professor, University of Cambridge
Other Study IDs: IRAS307166
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Vitiligo; Skin Abnormalities
MeSH Terms: conditions — Vitiligo; Skin Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Vitiligo
  Interventions: Device: Photoacoustic imaging
- Fitzpatrick Type 1
  Interventions: Device: Photoacoustic imaging
- Fitzpatrick Type 2
  Interventions: Device: Photoacoustic imaging
- Fitzpatrick Type 3
  Interventions: Device: Photoacoustic imaging
- Fitzpatrick Type 4
  Interventions: Device: Photoacoustic imaging
- Fitzpatrick Type 5
  Interventions: Device: Photoacoustic imaging
- Fitzpatrick Type 6
  Interventions: Device: Photoacoustic imaging

INTERVENTIONS:
Device: Photoacoustic imaging — Photoacoustic imaging

SUMMARY:
Photoacoustic imaging (PAI) is an emerging method which combines light and ultrasound to assess the blood content and oxygenation of the body. Light is absorbed by the blood, leading to the generation of ultrasound, from which the levels of oxygen can be derived. This high sensitivity to blood has seen it applied in multiple clinical trials for the assessment of a number of conditions including breast cancer assessment. However, the accuracy of the measurements and image quality is known to decrease as you look deeper into the body because light intensity decreases. Melanin in the skin is known to absorb light very strongly and so there is considerable concern that this may bias measurements made in people with darker skin tones compared to those with lighter skin tones. In this pilot study, we intend to recruit volunteers with a wide range of skin tones and vitiligo. We will scan a number of blood vessels and muscles using PAI and evaluate the photoacoustic measurements of blood content and oxygenation to identify, and ultimately correct for, biases in advance of further clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary adult non-vulnerable participants between the age of 20 to 70.
2. Can understand the Information sheet and give informed consent in English.
3. Normal or Overweight BMI (18.5 to 29.9)

Exclusion Criteria:

1. No participants who cannot give informed consent.
2. No tattoos or scarring of the regions to be imaged.
3. No pulmonary sleep disorder, or active respiratory disorders that may affect the blood oxygenation levels.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal adult population across range of skin tones
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Quantitative photoacoustic imaging | 1 year
  Identify biases in quantitative photoacoustic imaging when scanning people with different Fitzpatrick skin tones and Vitiligo.

IPD SHARING:
Plan to Share IPD: No